CLINICAL TRIAL: NCT06630377
Title: The Effectiveness of Galactooligosaccharide on the Treatment of Hyperuricemia
Brief Title: GOS and the Management of Hyperuricemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Min Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GOS-HUA-2024
Record Dates: First submitted 2024-07-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Subjects With Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention with GOS (Experimental): Eligible subjects are instructed to take one pocket of galactooligosaccharide during the first week, followed by two pockets of galactooligosaccharide during the remaining 7 weeks.
  Interventions: Dietary Supplement: GOS
- Dietary intervention with Placebo (Placebo Comparator): Eligible subjects are instructed to take one pocket of maltodextrin during the first week, followed by two pockets of maltodextrin during the remaining 7 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GOS — During the study period, subjects are instructed to take one pocket of galactooligosaccharide per day during the first week, followed by two pockets of galactooligosaccharide per day during the remaining 7 weeks. Aside from the dietary supplement provided, all participants are instructed to continue their normal routine and not make any changes to their dietary habits or physical activity.
  Arms: Dietary intervention with GOS
Dietary Supplement: Placebo — During the study period, subjects are instructed to take one pocket of placebo control per day during the first week, followed by two pockets of placebo control per day during the remaining 7 weeks. Aside from the dietary supplement provided, all participants are instructed to continue their normal routine and not make any changes to their dietary habits or physical activity.
  Arms: Dietary intervention with Placebo

SUMMARY:
Hyperuricemia is a major risk factor for many chronic diesease. Recently, gut mcirobiota has been identified as a novel therapeutic target for hyperuricemia. Both annimal studies and pilot human trials have demonstrated that administration of prebiotics help delay the progression of hyperuricemia throuh several mechanisms. This trial aims to examine the protective effects and potential mechanisms of galactooligosaccharide on hyperuricemia in clinical trials.

DETAILED DESCRIPTION:
Hyperuricemia is a major risk factor for many chronic diseases. Recently, dysbiosis of gut microbiota has been reported to play an important role in the pathogenesis of hyperuricemia. Animal studies have demonstrated that administration of prebiotics help delay the progression of hyperuricemia through several mechanisms such as reduction in endotoxemia, and enhanced production of short-chain fatty acids and hippuric acid.

However, whether administration of galactooligosaccharide also has a protective effect in subjects with hyperuricemia remain under-explored. Moreover, the molecular mechanisms underlying the protective effect of galactooligosaccharide remains largely unknown.

ELIGIBILITY:
Inclusion Criteria:

* Local residents aged between 18-80 years old;
* Stable weight (<5% weight change over the past 3 months);
* Fasting uric acid > 420 umol/L for male and > 360 umol/L for female on two different days;
* Not taking uric acid lowering drugs or have stopped taking uric acid lowering drugs for over 4 weeks at the time of recruitment;
* Absence of any diet or medication that might interfere with uric acid metabolism or gut microbiota, especially antibiotics, prebiotics or probiotics at the least 4 weeks before recruitment

Exclusion Criteria:

* Acute illness or evidence of any acute or chronic inflammatory of infective diseases;
* Participation in regular diet program more than 2 times per week in the latest 3 months prior to recruitment;
* Mental illness rendering them unable to understand the nature, scope, and possible consequences of the study;
* Women of childbearing age who are pregnant, breast-feeding or preparing for pregnancy; patients who had surgey within the past 6 months or planned surgery during the trial period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of serum uric acid | from baseline to 8 weeks after intervention
  change of serum uric acid level assessed by automatic biochemical detector
Change of excretion of uric acid | from baseline to 8 weeks after intervention
  excretion rate of uric acid assessed by secretion rate of uric acid in urine during 3 hours with automatic biochemical detector

SECONDARY OUTCOMES:
Change of gut microbiota | from baseline to 8 weeks after intervention
  Alterations of the composition of gut microbiota evaluated by metabogenomics and qPCR analysis in fecal samples with specific primers designed for each bacterium of interest
Change of microbial metabolites in the circulation | from baseline to 8 weeks after intervention
  Untargeted and targeted metabolomics will be used to assess the alterations of microbial metabolites in the circulation with high performance liquid chromatography-mass spectrometry with internal standards

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No